CLINICAL TRIAL: NCT01349387
Title: Effect of Treatment With Metformin in Type 2 Diabetes Patients on Alternative Genes Splicing Whose Maturation Depends on the Protein HuR, Including Gene Encoding Insulin Receptor
Brief Title: Effect of Treatment With Metformin in Type 2 Diabetes Patients on Alternative Genes Splicing
Acronym: METFORGENE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-A01389-30; 2011-000128-13 (EudraCT Number)
Record Dates: First submitted 2011-05-03; First posted 2011-05-06 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2011-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm1 (Experimental): During their visit of consultation on the follow-up to the type 2 diabetes, les patients will be selected on the basis of active metformin treatment at a dose greater than or equal to 1400 mg/day. Patients will have to achieve a 10 ml blood sample. The blood will be processed by Ficoll gradient centrifugation to remove the red cells and isolate circulating leukocytes: this stage will be conducted in the CERITD. Analysis on circulating leukocytes and in particular the quantification of expressions of isoforms A and B of the INSR1 by quantitative RT - PCR gene will be conducted in the laboratory of the Professor Marc Peschanski (unit INSERM 861 I - STEM of Evry).
  After inclusion in the study to J0, metformin treatment will be interrupted between J1 and J30, replaced by Januvia 100 mg/day dose, then resumed at J31.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — After inclusion in the study to J0, metformin treatment will be interrupted between J1 and J30, replaced by Januvia 100 mg/day dose, then resumed at J31.

SUMMARY:
Main objective : Show that treatment with metformin in patients with type 2 diabetes has an effect on alternative splicing of the insulin receptor.

Secondary objective : demonstrate that the effect on the ratio A/isoform B isoform with discontinuation of treatment with metformin can be réversé by the resumption of metformin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetic patients usually treated with metformin (≥ 1400 mg/day), associated or not to other oral anti-diabetic treatment or. injection treatment
* Patients major.
* Patients with a social security number
* Patients having signed a consent to participate in the study

Exclusion Criteria:

* Intolerance metformin
* Patients with type 1.
* Patients on pioglitazone or rosiglitazone
* Renal failure by an anomaly of the creatinine clearance (< 60 mL/min).
* Patients pregnant or likely to be.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Comparison of expression of isoforms A and B of the insulin receptor using quantitative RT PCR | inclusion (baseline), 30th days and 60th days
  comparison of the A isoform (without inclusion of exon 11) and B isoform (with inclusion of exon 11) ratio of the receptor in insulin, during the first period (without metformin) and the second period (with metformin)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CHARPENTIER, MD, Principal Investigator — CHSF-CERITD
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France